CLINICAL TRIAL: NCT05851014
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Trial of GB491 in Combination With Letrozole in Subjects With HR Positive and HER2 Negative Locally Advanced or Metastatic Breast Cancer Who Have Not Previously Received Systemic Therapy in This Disease Setting
Brief Title: A Study of GB491 in Combination With Letrozole in Patients With HR Positive and HER2 Negative Advanced Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GB491-008
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: HR+/HER2-; locally advanced or metastatic breast cancer; GB491
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB491 combined with Letrozole (Experimental)
  Interventions: Drug: GB491 combined with Letrozole
- Placebo combined with Letrozole (Placebo Comparator)
  Interventions: Drug: Placebo combined with Letrozole

INTERVENTIONS:
Drug: GB491 combined with Letrozole — Patients were randomized to receive GB491 150 mg orally twice daily, depending on their assignment. Letrozole 2.5 mg orally once a day from the first day of cycle 1 (one cycle every 28 days)
  Arms: GB491 combined with Letrozole
Drug: Placebo combined with Letrozole — Patients were randomized to receive placebo orally twice daily, depending on their assignment. Letrozole 2.5 mg orally once a day from the first day of cycle 1 (one cycle every 28 days)
  Arms: Placebo combined with Letrozole

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of GB491 combined with Letrozole versus placebo combined with Letrozole in the treatment of HR+/HER2- locally advanced or metastatic breast cancer without prior systemic antitumor therapy

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-75 years old;
* Have a pathologically-confirmed diagnosis of hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) breast cancer;
* No previous systematic antitumor therapy for locally advanced or metastatic breast cancer;
* Eastern Cooperative Oncology Group [ECOG] 0-1;
* Have adequate organ and marrow function;
* Agree to sign the informed consent;

Exclusion Criteria:

* Systematic treatment with any other CDK4/6 inhibitor；
* Subjects with known allergy to GB491 or any component of Letrozole；
* Confirmed diagnosis of HER2 positive disease;
* Known uncontrolled, or symptomatic central nervous system metastases;
* Had major surgery (or is expected to require major surgery during the study period), chemotherapy, radiation, any investigational drug, or other antitumor therapy within 4 weeks prior to randomization;
* Have previously received chemotherapy for locoregionally recurrent or metastatic breast cancer;
* Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure, or ventricular arrhythmia which need medical intervention；
* Known history of HIV infection or HIV seropositivity (including HIV antibody positive at the time of screening)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed PFS based on RECIST v1.1 | Approximately 60 months
  To evaluate progression-free survival (PFS) of GB491 plus Letrozole versus placebo plus Letrozole in HR+/HER2- locally advanced or metastatic breast cancer without prior systemic antitumor therapy (as assessed by the investigator).

SECONDARY OUTCOMES:
BICR-assessed PFS based on RECIST v1.1. | Approximately 60 months
OS | Approximately 60 months
ORR | Approximately 60 months
DOR | Approximately 60 months
DCR | Approximately 60 months
CBR | Approximately 60 months
Number of Participants With adverse events (AEs) and serious adverse events (SAEs) Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0 | Approximately 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Ph.D, Principal Investigator — Fudan University
Locations (52):
- China (52):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Hospital of Anhui Medical University, Hefei, Anhui
  - Anhui Cancer Hospital, Hefei, Anhui
  - The Second Hosptial of Anhui Medical University, Hefei, Anhui
  - Betjing Tiantan Hosptial，Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospial, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of Wenzhou Medical University, Wenzhou, Fujian
  - The First Affiliated Hosptial of Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-Sen University Cancer Center(Huangpu Campus), Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center(Yuexiu Campus), Guangzhou, Guangdong
  - Maternal and Child Healh Hosptal of Guangdong Provrce, Guangzhou, Guangdong
  - Meizhou People's Hosptial, Meizhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hosptial of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First Affiliated Hosptial of Nanchang University, Nanchang, Jiangxi
  - The Nanchang theird people's Hosptial, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shangrao People's Hospital, Shangrao, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yingchuan, Ningxia
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hosptial of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - First Hosptial of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuang University, Chengdu, Sichuang
  - Tianjin Mediacl University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Cancer Affiliated Hospital of Xingjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hosptial, Kunming, Yunnan
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No